CLINICAL TRIAL: NCT05318222
Title: Virtual Platforms for Genetics Evaluation in the Medically Underserved
Brief Title: Genetic Inclusion by Virtual Evaluation
Acronym: GIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Seema Lalani, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-50430
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Birth Defects; Multiple Congenital Anomaly; Neurodevelopmental Disorders
MeSH Terms: conditions — Congenital Abnormalities; Abnormalities, Multiple; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WGS arm (Other): All 200 patients recruited will undergo WGS
  Interventions: Diagnostic Test: Whole genome sequencing (WGS)

INTERVENTIONS:
Diagnostic Test: Whole genome sequencing (WGS) — WGS will identify copy number variations (CNVs), single nucleotide variants (SNVs), as well as triplet repeat disorders in children with rare diseases

SUMMARY:
This study aims to transform the current clinical practice paradigm by leveraging an internally designed web-based model of delivery of care called Consultagene to provide remote evaluation and genomic sequencing for improving genetic health of less resourced children with rare disorders living along the Texas-Mexico border.

DETAILED DESCRIPTION:
Inadequate access to genetics evaluation and genomic testing in the Hispanic minorities living along the Texas-Mexico has marginalized the most vulnerable pediatric group. In this study, we will (1) implement a virtual web-based service, called Consultagene for simplifying patient pathways and deliver virtual genetics evaluation in Rio Grande Valley (RGV) (2) provide rapid genetic diagnoses through whole genome sequencing and interpretation of diagnostic studies for medical decision-making and improving health outcomes for the minorities, and (3) build genomic competency of front-line healthcare providers through education and machine learning to expedite referral of pediatric patients with suspected rare diseases for shortening diagnostic odyssey.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patients with undiagnosed rare genetic diseases residing in the Rio Grande Valley and El Paso in Texas

Exclusion Criteria:

Children with known genetic diseases

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seema Lalani, Principal Investigator — Baylor College of Medicine
Locations (1):
- University of Texas Rio Grande Valley, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No